CLINICAL TRIAL: NCT06759935
Title: Randomized, Sham Controlled, Single Blind Study on the Performance and Safety of Photo Biomodulation Therapy (PBMT) With LightForce® Therapy Lasers on Shoulder Soft Tissue Inflammation Pain Reduction
Brief Title: Performance and Safety of LightForce® Therapy Lasers on Shoulder Soft Tissue Inflammation Pain Reduction
Acronym: SHINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DJO UK Ltd (Industry)
Collaborators: Donawa Lifescience Consulting (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENOVIS-S-INP-0010
Record Dates: First submitted 2024-12-23; First posted 2025-01-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome; Rotator Cuff Tendinitis
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome; Rotator Cuff Injuries | interventions — Laser Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Laser treatment - Arm 1 (Sham Comparator): Sham Laser therapy
  Interventions: Device: Sham Laser therapy; Other: physiotherapy/exercise protocol
- Laser Treatment - Arm 2 (Active Comparator): Laser therapy
  Interventions: Device: Laser therapy; Other: physiotherapy/exercise protocol

INTERVENTIONS:
Device: Sham Laser therapy — sham laser therapy for 4 consecutive weeks with a minimum of 3 sessions per week.
  Arms: Sham Laser treatment - Arm 1
Device: Laser therapy — laser therapy for 4 consecutive weeks with a minimum of 3 sessions per week.
  Arms: Laser Treatment - Arm 2
Other: physiotherapy/exercise protocol — physiotherapy/exercise protocol represents the standard of care (SOC) and the program includes Codman's pendulum exercise, range of motion (ROM) exercises, stretching and isometric strengthening exercises, for 4 consecutive weeks with a minimum of 3 sessions per week.

SUMMARY:
DJO UK Ltd (ENOVIS) is conducting this study to assess the effectiveness of LightForce® Therapy Lasers on pain reduction in shoulder soft tissue inflammation. In detail this study will assess superiority of LightForce® Therapy Lasers combined with standard of care, represented by physiotherapy/exercise program compared to sham laser combined with standard of care (physiotherapy/exercise program) on pain reduction in subjects with shoulder soft tissue inflammation due to Impingement (Subacromial impingement syndrome (SAIS)) or Rotator Cuff Tendinopathy (RCT),. In addition, this study allows to collect post market clinical data on the safety and performance of LightForce® Therapy Lasers, when used, following the normal clinical practice, in accordance with its approved and CE marked intended use.

DETAILED DESCRIPTION:
This clinical investigation is a post-market, International, multi center, prospective, randomized, sham controlled, single blind study to assess the effectiveness of LightForce® Therapy Lasers and to collect PMCF data on the safety and performance of LightForce® Therapy Lasers, when used in accordance with its approved labeling, to comply with Medical Device Regulation (EU) 2017/745 (MDR) Article 61 and Part B of Annex XI.

ELIGIBILITY:
Inclusion Criteria:

1. Patient male or female with age ≥18 years old
2. Patient with diagnosis of shoulder soft tissue inflammation due to SAIS/RCT (as confirmed by physical examination and/or imaging) to be treated by LightForce® Therapy Lasers according to its indications.
3. Patient suffering from shoulder soft tissue inflammation due to SAIS/RCT pain for more than 3 months prior to enrollment
4. Pain (either persistent or during activities) score reported by the subject at baseline ≥ 40 mm measured on VAS
5. Patient able to provide written informed consent

Exclusion Criteria:

1. Patient with musculoskeletal pathological conditions not to be treated with/contraindication to the use of LightForce® Therapy Lasers according to its intended use and indications
2. Patients who are taking drugs that have heat or light sensitive contraindications, such as but not limited to certain types of steroids
3. Patients who are administered with corticosteroids, should discontinue the treatment at least 2 weeks prior to study treatment start
4. Pregnant females or females of childbearing potentially planning to become pregnant during the study participation
5. Patients who had systemic inflammatory conditions (i.e.rheumatoid arthritis, polymyalgia rheumatica)
6. Patients who underwent intra-articular injection (Ialuronic acid, platelet rich plasma or corticosteroids) in the shoulder in the last 3 months
7. Patients who have a disease that would limit their participation in exercises (i.e. severe chronic obstructive pulmonary disease, severe heart failure, cerebrovascular event history)
8. Patients with a prior history of surgical intervention and implantation of a metal implant into the affected shoulder
9. Patients with a diagnosis of active cancer
10. Patients with tattoos covering more than 30% of the area to be treated with LightForce® Therapy Lasers
11. Patients who are mentally or physically incapacitated
12. Patient participating in other clinical study or has completed a clinical study less than 30 days prior to enrollment
13. Patient affected by shoulder soft tissue acute inflammation due to recent sport injury or trauma
14. Patients with other musculoskeletal problems of the shoulder joint such as calcifying tendinitis, full thickness rotator-cuff tear, adhesive capsulitis, fibromyalgia, recent surgery or fracture of the shoulder joint, and/or undergoing to specific physiotherapy for these ("recent" is defined as within 30 days prior to enrollment).
15. Patients with other clinically significant co-morbidities that make the patient unsuitable for study participation, at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain change | 4 weeks after treatment start
  Pain reduction measured with Visual Analog Scale (VAS) (in a scale 0-100 mm, where 0 is no pain and 100 is the worst possible pain) after 4 weeks of treatment compared to pre-treatment (baseline) VAS

SECONDARY OUTCOMES:
Safety - adverse event rate | through study completion, an average of 21 weeks
  Proportion of patient experiencing an adverse event associated with device use

OTHER OUTCOMES:
Pain change | 1,2,3,6, 9 and 12 weeks
  Pain measured with Visual Analog Scale (VAS) (in a scale 0-100 mm, where 0 is no pain and 100 is the worst possible pain) at 1,2,3,6, 9 and 12 weeks after treatment start to assess short-term and long-term pain management compared to baseline
Shoulder pain and disability | 2, 4, 6 and at 12 weeks
  Shoulder pain and disability measured with the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire (the score output is given as a percentace -from 0% to 100%- and the lower the percentage the better is the clinical outome, the higher the percentage the worse is the clinical outcome) performed at 2, 4, 6 and at 12 weeks after treatment start compared to baseline.
Patient overall status change | 2, 4, 6 ans 12 weeks after treatment start
  Patient ratings of overall improvement, assessed by QoL (SF-12): The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. The SF-12 uses 12 items and scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. SF-12 will be assessed at 2, 4, 6 weeks and at 12 weeks and compared to baseline
Range of motion (ROM) for shoulder | 2, 4, 6 ans 12 weeks after treatment start
  Range of motion for shoulder both passive and active, pain free and at maximum ROM, in all the planes of motion, measured by a universal goniometer at2, 4, 6 ans 12 weeks after treatment start compared to baseline
Neer test | 2, 4, 6 ans 12 weeks after treatment start
  Functional test to assess shoulder pain onset at a certain degree of movement during flexion and pressure application (often used as a diagnositc tool of subacromial impingement) performed at 2,4, 6 and at 12 weeks after treatment start and compared to baseline
Palm up test | 2, 4, 6 ans 12 weeks after treatment start
  Functional test where the patient elevates the extended arm with the palm facing upwards and against examiner's resistance, presence of pain can denote tendonitis (often used as diagnostic tool) and performed at 2,4, 6 and at 12 weeks after treatment start and compared to baseline
Jobe test | 2, 4, 6 ans 12 weeks after treatment start
  Functional testing of the arm with the thumb in 'thumbs up' and resistance provided by the examiner, weakness or pain would represent a positive test indicating a tear of the supraspinatus muscle or tendon, it will be performed at 2,4, 6 and at 12 weeks after treatment start and compared to baseline
Pain change | 18 weeks after treatment start
  pain measured with Visual Analog Scale (VAS) (in a scale 0-100 mm, where 0 is no pain and 100 is the worst possible pain) to assess post study pain
Rate of patients needed new treatment | 18 weeks after treatment start
  Patients will be asked through a questionnaire whether any new treatment and in case which one (pharmacological, physiotherapic etc) was needed to manage shoulder pain after 12 weeks from treatment start

CONTACTS AND LOCATIONS:
Overall Officials: ANDREA TURIACO, Physiotherapist, Principal Investigator — Fisioterapia Gardenie
Locations (10):
- Cabinet Attal, Serris, France
- Italy (6):
  - Fisioterapia Carioni, Cassano d'Adda, Milano
  - Casertafisio, Caserta
  - Rachis Center, Roma
  - Fisiolab3, Roma
  - Fisioterapia Eur, Roma
  - Fisioterapia Gardenie, Roma
- United Kingdom (3):
  - Freedom Care Clinics, Leeds
  - Indergaard Physiotherapy Ltd, Leeds
  - Freedom Care Clinic, Manchester

IPD SHARING:
Plan to Share IPD: No